CLINICAL TRIAL: NCT05914857
Title: Evaluation of the Safety and Efficacy of SGLT2 Inhibitors in Pre-diabetic Patients: A Randomized Trial
Brief Title: Evaluation of the Safety and Efficacy of SGLT2 Inhibitors in Pre-diabetic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangjin (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor-Investigator, Yangjin, Associate chief physician, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 80497
Record Dates: First submitted 2023-05-06; First posted 2023-06-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Prediabetic State; Impaired Fasting Glucose; Impaired Glucose Tolerance
Keywords: Prediabetic State; Impaired Fasting Glucose; Impaired Glucose Tolerance; Sodium-glucose co-transporter 2 inhibitor; Dapagaliflozin
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will be administered Dapagliflozin 10 mg/day in addition to lifestyle intervention.
  Interventions: Drug: Dapagliflozin 10mg Tab; Behavioral: lifestyle interventions
- Control group (Placebo Comparator): Patients in the control group will be given lifestyle intervention only.
  Interventions: Behavioral: lifestyle interventions

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin Tablets, Oral, 10mg, Once daily
  Other Names: Dapagliflozin Tablets
  Arms: Intervention group
Behavioral: lifestyle interventions — Consisting of 30 minutes of moderate-intensity exercise every day and a reduction of 300 calories in the total diet

SUMMARY:
Pre-diabetes is a state characterized by subclinical impairment in glycemic variables that is intermediate between normal glucose tolerance (NGT) and diabetes. There are two frequently used definitions for pre-diabetes, one from the American Diabetes Association (ADA) and another from the World Health Organization (WHO), and both include impaired glucose tolerance (IGT), impaired fasting glucose (IFG), and a calibrated hemoglobin A1c (HbA1c) of between 5.7 and 6.4%. More than 30 % of the global population demonstrated one or more forms of prediabetic dysglycaemia. In general, approximately 70 % of individuals with IFG and/or IGT can expect to go on to develop clinical type 2 diabetes at some time in the future, and the risk increases with higher HbA1c levels and with higher BMI. Worse still, the prevalence of pre-diabetes is increasing worldwide, with a growing number of patients progressing to diabetes. Identification and treatment of pre-diabetic individuals is therefore crucial. Recent evidence suggested that preventing progression of pre-diabetes to diabetes is possible, and thus efficacious interventions for pre-diabetic individuals are the cornerstone of diabetes prevention.

The current paradigm for diabetes prevention in high-risk individuals focuses on achieving moderate weight loss via dietary change and increasing physical activity. However, lifestyle-based weight-loss strategies may initially be successful, but difficult to achieve or maintain.

In many cases, pharmacologic treatments may be needed to regulate blood glucose. Randomized clinical trials (RCTs) have verified the efficacy of metformin in preventing insulin resistance syndrome, along with the progression of microvascular diseases and heart attacks. Meanwhile, clinical experience and trial data have yielded almost no significant safety concerns for metformin. Nonetheless, it may cause discomfort for up to 25% of patients who experience diarrhea and nausea subsequent to its administration. For patients with a contraindication or intolerable adverse effects to metformin, Sodium Glucose Cotransporter 2 (SGLT-2) inhibitors with novel mode of action may be another alternative.

Large clinical trials have not yet identified a substantial elevation in the frequency of adverse reactions related to SGLT-2 inhibitors when compared to the placebo group. Inhibition of SGLT-2 has some extra advantages for diabetes management over other therapeutic approaches. Firstly, the SGLT-2 is exclusively expressed in renal proximal tubules, and thus selective inhibitors will exert a glucose-lowering effect, independently of insulin secretion. Therefore, SGLT-2 inhibitors can cause weight loss without inducing major hypoglycemic events. Secondly, the cardiovascular benefits of SGLT-2 inhibitors was supported by large clinical trials in the modern context of antiplatelet, statin, and blood pressure management, which may match many of the advantages of metformin. Thirdly, SGLT-2 inhibitors have also been proven to prevent nephropathy for its restriction on albuminuria and inflammatory processes, and to subsequently dampen the deterioration in renal function. Overall, SGLT-2 inhibitors have demonstrated safety in non-diabetic patients, particularly in those afflicted with heart or kidney failure, and have shown to provide additional benefits.

At present, the overall effectiveness and safety of SGLT-2 inhibitors in improving metabolism of pre-diabetic patients are still unclear. The purpose of this experiment is to evaluate the effect of SGLT-2 inhibitor on pre-diabetic patients.

DETAILED DESCRIPTION:
1. Study design

   This study is a prospective, single-center parallel-group trial conducted at the Third Hospital of Peking University. Pre-diabetic patients will be included in the study if they meet the inclusion and exclusion criteria. The participants will be stratified by gender (male: female =1:1) and then randomly allocated to the intervention and control groups using a random number table. Patients in the intervention group will be administered Dapagliflozin 10 mg/day in addition to lifestyle intervention, while patients in the control group will be given lifestyle intervention only. Recommended lifestyle interventions include 30 minutes of moderate intensity exercise per day, with a total calorie reduction of 300 calories, according to Intervention for Adults with Pre-diabetes: A Chinese Expert Consensus.

   The specific goals of lifestyle intervention include achieving or approaching a BMI of 24 kg/m2 for overweight or obese individuals, or at least a 5% initial weight loss within 3-6 months. Patients should not initiate during the study an organized diet and/or exercise weight reduction program other than the lifestyle and dietary measures for diabetes treatment. Study participants should be instructed not to donate blood or blood products during the study.

   Physical activity: For optimal physical fitness, it is highly recommended to incorporate a combination of aerobic and resistance exercises daily for a minimum of 30 minutes. Aerobic exercises, including brisk walking, jogging, cycling, and swimming, should be performed at least three times weekly. Resistance exercises, which entail the utilization of resistance training equipment or free weights (such as dumbbells and barbells), should be integrated into the exercise regimen at least twice a week, in conjunction with regular aerobic exercise.

   Dietary intervention: It is recommended that the daily total energy requirement comprises of 45%-60% from carbohydrates, 25%-35% from fats, and 15%-20% from protein. Additionally, it is advised that the daily dietary energy intake be reduced by a minimum of 300 kCal. Furthermore, it is crucial to limit the intake of saturated fatty acids to less than 30% of the total fat intake, and restrict daily salt intake to no more than 6g. Lastly, it is not advisable to consume alcohol, or if consumed, it must be included in the total energy intake.

   A sample size estimation is implemented for this trial based on the comparison of the intervention and control groups with respect to the primary efficacy end point, the change from baseline at 12 weeks in 2h plasma glucose on an oral glucose tolerance test (OGTT) (2h-PG). The estimated decrease of 2hPG in the intervention and the control group is 2% and 1%, respectively. Additionally, participants will be stratified according to gender, as one purpose of this study is to explore whether and to what extent the drug has adverse effects on various genitourinary system. After a careful search of the relevant literature, the ratio of male to female pre-diabetic patients is approximately 1:1. Therefore, under the assumption of an estimated 10% dropout rate at 12 weeks in this trial, a total sample size of 120 participants, including 30 participants allocating to the intervention group and 30 participants to the control group in each gender, will provide the trial with 80% power to demonstrate the superiority of treatment with the use of a two-sample t-test at a two-sided alpha level of 0.05. Previous studies have indicated that approximately 30% of patients are over the age of 50, so it is anticipated to include:

   A. 42 males under 50 years old B. 18 men aged 50-65. C. 42 women under 50 years old. D. 18 women aged 50-65.
2. Research process 1) Screening period. Individuals who meet the inclusion criteria and demonstrate good adherence to medication regimens will be eligible for inclusion in the study, and will be randomly assigned to the intervention and control groups. Subsequently, their basic information will be collected, including age, sex, body mass index (BMI), blood pressure, abdominal circumference, smoking history, cardiovascular disease history, amputation history, use of hypoglycemic and/or slimming drugs, history of biochemical hypoglycemia serious liver disease history, malignant tumor history, stroke history, and urogenital infection history. Then participants will undergo serial blood and urine testing for blood glucose and other metabolism parameters. Male participants may also receive semen analysis voluntarily. Finally, patients in the intervention group will be administered Dapagliflozin 10 mg/day in addition to lifestyle intervention, while patients in the control group will be only given lifestyle intervention.

2) Follow-up stage. The follow-up cycle will be computed subsequent to the initiation of the intervention. Telephone follow-up will be carried out at week 4 and week 8 to assess the subjects' adherence to the prescribed medication, evaluate any potential adverse drug reactions, and record the type and time of physical activities. Concurrently, we will conduct patient education, optimize their treatment plans, and collect the incidence of pregnancy. Corresponding data will be recorded on the case report form.

During the final visit, clinical information of the participants will be obtained, including body mass index (BMI), blood pressure (BP), and waist circumference (WC). For female participants, pregnancy will be confirmed. In addition, serial blood and urine tests will be performed to examine blood glucose and other metabolic parameters. Finally, a summary of the experiment's process will be documented.

3.Statistical analysis We will utilize SPSS 25.0 software for statistical analysis. All statistical tests are two-tailed tests, and a P value of less than or equal to 0.05 will be considered statistically significant. Continuous data will be presented as mean ± SD if the measurement data are normally distributed. An independent sample t-test will be used to compare the different therapeutic effects between the parameters with and without the intervention of SGLT-2 inhibitors. Counting data will be represented as medians and interquartile ranges [IQRs], and compared using a Chi-square test between groups. Spearman's correlation analysis and binary logistic regression analysis will be employed for correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 ~65 years old;
2. OGTT received within half a year and were diagnosed with prediabetes In accordance with the gout classification criteria of the American Diabetes Association: ① Fasting blood glucose (FPG)≥6.1 mmol/L and < 7.0 mmol/L; ② The blood glucose (2h-PG) concentration at OGTT 2h was ≥7.8 and < 11.1mmol/L; ③ Glycosylated hemoglobin (HbA1c) ≥5.7% and < 6.4%;
3. No antidiabetic drugs (including traditional Chinese medicine) were taken within 6 months before screening;
4. Sign the informed consent form.

Exclusion Criteria:

1. Diagnosed with diabetes;
2. Taking medications that affect glucose and lipid metabolism (excluding thiazide diuretics at a daily dose of ≤ 12.5 mg);
3. Taking weight-loss drugs (including traditional Chinese medicine) within 6 months before screening;
4. Patients with acute infection, surgery, acute alcoholism, mental illness, etc;
5. Patients with liver and kidney dysfunction, severe chronic gastrointestinal disease, uncontrolled thyroid disease, cancer, and ventilator use;
6. Systolic blood pressure ≥180 mmHg (1 mmHg = 0.133 kPa) or diastolic blood pressure ≥110 mmHg at screening;
7. Electrocardiogram within 12 weeks before screening indicating arrhythmia requiring urgent diagnosis or treatment (e.g., clinically newly identified severe arrhythmia or conduction disturbance), myocardial infarction, unstable angina, or stroke requiring cardiovascular and cerebrovascular intervention;
8. A history of traumatic amputation within the past year, or active skin ulcers, osteomyelitis, gangrene, or critical lower limb ischemia within the past 6 months;
9. Enrolled in drug/device clinical studies (including vaccines) within 12 weeks before screening;
10. Pregnant, lactating women, or those planning a recent pregnancy;
11. Allergic constitution or multi-drug allergy;
12. Receiving bariatric surgery within the past 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
2h plasma glucose on an oral glucose tolerance test (OGTT) | Change from baseline (time 0) to study end (12 weeks)
  2h-PG change

SECONDARY OUTCOMES:
Change in HbA1c | Change from baseline (time 0) to study end (12 weeks)
  fasting serum HbA1c change
Change in Body Weight | Change from baseline (time 0) to study end (12 weeks)
  fasting body weight change
Change in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) | Change from baseline (time 0) to study end (12 weeks)
  Change in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Change in Waist Circumference (WC) | Change from baseline (time 0) to study end (12 weeks)
  Change in Waist Circumference (WC)
Glycemic control including Fasting Blood Glucose (FBG) and Glycosylated Hemoglobin (HbA1C) | Change from baseline (time 0) to study end (12 weeks)
  Glycemic control including Fasting Blood Glucose (FBG) and Glycosylated
Plasma lipid fractions including Total Cholesterol Levels (CHOL) and Triglyceride (TRG) Levels | Change from baseline (time 0) to study end (12 weeks)
  Plasma lipid fractions including Total Cholesterol Levels (CHOL) and Triglyceride
Liver Enzymes including ALT and AST levels | Change from baseline (time 0) to study end (12 weeks)
  Liver Enzymes including ALT and AST levels
Creatinine, calculated eGFR, and Albumin/Creatinine Ratio (ACR) | Change from baseline (time 0) to study end (12 weeks)
  Creatinine, calculated eGFR, and Albumin/Creatinine Ratio (ACR)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, doctorate, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Xia L, Yin D, Yang J, Wei R. Evaluating the Safety and Efficacy of Sodium-Glucose Co-transporter 2 Inhibitors in Subjects with Prediabetes: A Protocol for a Randomized Controlled Trial. Diabetes Ther. 2024 May;15(5):1231-1244. doi: 10.1007/s13300-024-01560-3. Epub 2024 Mar 18. PMID 38494571